CLINICAL TRIAL: NCT06091384
Title: The Effects of Based-home High-resistance Inspiratory Muscle Training on Neurovascular Control, Blood Pressure, and Exercise Capacity in Patients With Post-COVID-19 Syndrome
Brief Title: Inspiratory Muscle Strength Training in Post-Covid Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: D'Or Institute for Research and Education (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IMST
Record Dates: First submitted 2023-10-17; First posted 2023-10-19 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Cardiovascular Abnormalities; Post-COVID-19 Syndrome; Physical Exercise
MeSH Terms: conditions — Cardiovascular Abnormalities; Post-Acute COVID-19 Syndrome; Motor Activity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inspiratory Muscle Strength Training (Experimental): Using a handheld device, participants will perform 30 breaths a day at 75% of maximal inspiratory pressure, six days a week, for 6 weeks.
  Interventions: Other: Inspiratory muscle strength training
- Sham- Inspiratory Muscle Training (Sham Comparator): Using a handheld device, participants will perform 30 breaths a day at 15% of maximal inspiratory pressure, six days a week, for 6 weeks.
  Interventions: Other: Inspiratory muscle strength training

INTERVENTIONS:
Other: Inspiratory muscle strength training — Using a handheld device, participants will perform 30 breaths per day at 75% of maximal inspiratory pressure, six days a week, during 6 weeks.

SUMMARY:
Patients with post-Covid-19 syndrome are at high risk of developing cardiovascular diseases 12 months after acute infection of COVID-19. We recently revealed that these patients have elevated muscular sympathetic nerve activity (MSNA), vascular dysfunction, impaired cardiac diastolic function, and reduced functional capacity. Considering that these outcomes are independent predictors of cardiovascular mortality, it is urgent to restore the cardiovascular health of these patients. High resistance inspiratory muscle strength training (IMST) at 75% of pressure inspiratory (PImax) performed at home (5 min/session, 5-7 times/week per 6 weeks) reduces the MSNA, improves the endothelial function and lowers blood pressure in different populations. Based on these findings, IMST (75% PImax) is an excellent therapeutic option for patients with post-COVID-19 syndrome. Therefore, the aim of the present proposal is to test whether IMST (75% PImax) reduces sympathetic activity, improves vascular function, and restores cardiac function, evoking an increase in functional capacity in patients with post-COVID-19 syndrome. To test these hypotheses we will conduct a randomized, double-blind, sham-controlled clinical trial to test these hypotheses.

ELIGIBILITY:
Inclusion Criteria:

* Post-COVID-19 syndrome
* Have been diagnosed with COVID-19 by RT-PCR
* Have oxygen saturation ≤ 93% in room air during the acute phase of the COVID-19
* Have received oxygen supply from any device during the acute phase of the COVID-19
* Hospitalization to treat the Covid-19
* Participants in cardiopulmonary rehabilitation or physical conditioning programs

Exclusion Criteria:

* Pregnant
* History of chronic obstructive pulmonary disease or dependence on oxygen support
* History of cardiovascular and renal diseases and cancer prior to the COVID-19 diagnosis
* Difficulties in moving to the laboratory for assessments

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-10-16 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
Muscle sympathetic nerve activity | Baseline and 6 weeks after ISMT and Sham
  Microneurography
Endothelial function | Baseline and 6 weeks after ISMT and Sham
  Doppler Ultrasound
Arterial stiffness | Baseline and 6 weeks after ISMT and Sham
  Applanation tonometry
Blood pressure | Baseline and 6 weeks after ISMT and Sham
  Sphygmomanometry
Exercise Capacity | Baseline and 6 weeks after ISMT and Sham
  Cardiopulmonary exercise testing
Maximum inspiratory pressure | Baseline and 6 weeks after ISMT and Sham
  Manovacuometry

SECONDARY OUTCOMES:
Oxidative stress | Baseline and 6 weeks after ISMT and Sham
  Blood samples
Nitric oxide | Baseline and 6 weeks after ISMT and Sham
  Blood samples
Inflammatory profile | Baseline and 6 weeks after ISMT and Sham
  Blood samples

CONTACTS AND LOCATIONS:
Locations (1):
- D'Or Institute of Research and Education, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No